CLINICAL TRIAL: NCT05942976
Title: Ultrasonographic Differences in Entheses in Rheumatoid Arthritis and Axial Spondyloarthropathy Patients
Brief Title: Enthesis Differences in Rheumatoid Arthritis and Axial Spondyloarthropathy
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Tayyip Dede, Medical Doctor, Istanbul Training and Research Hospital
Other Study IDs: 16/09/2022; 2011-KAEK-50;288
Record Dates: First submitted 2023-06-27; First posted 2023-07-12 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Axial Spondyloarthritis; Rheumatoid Arthritis; Enthesitis; Enthesopathy
Keywords: Axial Spondyloarthritis,; Rheumatoid Arthritis; Enthesitis; Ultrasound
MeSH Terms: conditions — Axial Spondyloarthritis; Arthritis, Rheumatoid; Enthesopathy | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: axial spondyloarthritis: SpA patients identified according to the Assessment of Spondyloarthritis classification criteria
  Interventions: Other: ULTRASOUND
- group 2: Rheumatoid arthritis: RA patients identified according to the 2010 American College of Rheumatology/Europan Leage Against Rheumatism classification criteria
  Interventions: Other: ULTRASOUND
- group:3 Healthy Control: healthy controls with no history of rheumatic diseases
  Interventions: Other: ULTRASOUND

INTERVENTIONS:
Other: ULTRASOUND — 10 enthesis areas will be evaluated in 20 minutes with ultrasound.

SUMMARY:
The aim of this study is to investigate the sonographic differences in entheses in patients with Rheumatoid arthritis and Axial Spondyloarthropathy.

DETAILED DESCRIPTION:
After recording the demographic data of the patients; 5 enthesis regions 5 enthesis sites were evaluated bilaterally as ''tricipital tendon (TT), quadricipital tendon (QT), proximal patellar tendon (PPT), distal patellar tendon (DPT), achilles tendon (AT)'' will be sonographically evaluated and the presence of hypoechogenicity , tendon thickness increase, power Doppler activity, erosion, presence of entezophyte/calcification will be investigated. The differences between the groups will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients identified according to the 2010 American College of Rheumatology /Europan Leage Against Rheumatism classification criteria,
* axial Spondyloarthrtis patients identified according to the Assessment of Spondyloarthritis classification criteria
* healthy controls with no history of rheumatic diseases.

Exclusion Criteria:

* history of limb trauma and surgery in the last 3 months,
* metabolic disease (diabetes mellitus, hypothyroidism),
* malignant neoplasm,
* limitation of range of motion in the extremity,
* those who have received corticosteroid injections in the last 3 months,
* uncontrollable fibromyalgia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients identified according to the 2010 American College of Rheumatology /Europan Leage Against Rheumatism classification criteria, axial Spondyloarthrtis patients identified according to the Assessment of Spondyloarthritis classification criteria and healthy controls with no history of rheumatic diseases.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Ultrasound enthesis differences between the groups | 2 months
  triceps tendon, quadriceps tendon, proximal patellar tendon, distal patellar tendon and achilles tendons enthesitis scores differences between the groups
The relationship between ultrasound findings and disease parameters | 2 months
  The relationship between triceps tendon, quadriceps tendon, proximal patellar tendon, distal patellar tendon and achilles tendons enthesitis scores and Clinical disease activity index and BASDAI

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Resarch Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes